CLINICAL TRIAL: NCT05400473
Title: Effects of Adding Photobiomodulation to a Specific Therapeutic Exercise Program for the Treatment of Individuals With Chronic Nonspecific Neck Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cid André Fidelis de Paula Gomes (Other)
Responsible Party: Sponsor-Investigator, Cid André Fidelis de Paula Gomes, Phd, professor, University of Nove de Julho
Organization: University of Nove de Julho (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 58616022.1.0000.5511
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Neck Pain; Chronic Pain
MeSH Terms: conditions — Neck Pain; Chronic Pain | interventions — Exercise Therapy; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigator will not be part of any assessment or treatment process.
  Two researchers will be solely responsible for evaluating the outcomes. These will not participate in any other process. And they did not know the allocation of participants in their respective groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic exercise group (Active Comparator): 1.Movements of flexion, extension, inclinations, and rotations of the cervical region at maximum amplitude and without load. 2.Neural mobilization of the cervical nerve roots. 3.Contraction of the deep muscles of the flexors, extensors, and rotators of the cervical region without performing spinal movements, using the movement of the eyes to aid in the accomplishment of these exercises. 4.Isometric contraction of the flexor muscles, inclinators, and rotators against manual resistance of the physiotherapist. 5.Isometric contraction of the cervical extensors of the cervical region against gravity. 6.Contraction of the flexor muscles, extensors, and incliners of the cervical region against the resistance of elastic bands.
  Interventions: Other: Therapeutic exercise
- Therapeutic exercise group + photobiomodulation (Experimental): This group will consist of 30 participants. Initially, photobiomodulation will be applied on the cervical region. A low-power infrared laser therapy unit (Therapy XT - ANVISA RDC Standard 185/2001 - DMC, São Paulo, SP, Brazil) will be used to carry out the photobiomodulation protocol. The infrared laser therapy unit to be used has the characteristics: continuous optical output of 100 mW, with a wavelength of 808 nm, beam size area of 0.028 cm2, power density 1.78 W/cm2, with 7 Joules per point, with a duration of 70 seconds of application for each point.For application, the individual will be seated. With the cervical region bare, the therapist will position the tip of the laser therapy unit perpendicularly on each of the 12 predefined points along the cervical region (6 points laterally to the right and 6 points laterally to the left).
  Interventions: Other: Therapeutic exercise; Other: Photobiomodulation

INTERVENTIONS:
Other: Therapeutic exercise — This group will consist of 30 participants. A program consisting of specific therapeutic exercises for the cervical region will be applied.
Other: Photobiomodulation — Photobiomodulation will be applied on the cervical region. To perform the photobiomodulation protocol, a low power infrared laser therapy unit will be used.
  Arms: Therapeutic exercise group + photobiomodulation

SUMMARY:
In the current clinical and scientific reality, conservative treatment is the most coherent clinical management with a view to the proper rehabilitation of patients with chronic neck pain, with a trend towards the use of therapeutic exercise. However, some uncertainty about the effectiveness of therapeutic exercises still remains, requiring further studies with high methodological rigor, especially with regard to multimodal treatment, such as the combination of therapeutic exercises with photobiomodulation. Thus, the objective of this project is to evaluate the effects of adding photobiomodulation to a program of specific therapeutic exercises for the treatment of individuals with chronic non-specific neck pain. For this, 60 participants will be randomized into two groups: therapeutic exercise group + photobiomodulation (n = 30), and therapeutic exercise group (n = 30). There will be 10 treatment sessions and participants will be evaluated before, after the 10 sessions, and 4 weeks after the end of treatment using the Numerical Pain Scale, Neck Disability Index, Catastrophic Thoughts about Pain Scale, and Tampa Kinesiophobia Scale. In the statistical analysis, a linear mixed model will be applied, considering the interaction between the time and group factors. Finally, the addition of photobiomodulation to a therapeutic exercise program is expected to generate clinical improvements for patients with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* With chronic neck pain (for more than 90 days)
* Identified according to the following criteria: NDI score ≥ 5
* Numerical Pain Scale (END) score ≥ 3 at rest or during active neck movement

Exclusion Criteria:

* Individuals who had a history of cervical trauma; head, face, or cervical surgery
* Degenerative diseases of the spine
* Pain radiating to the upper limbs
* Having been submitted to physiotherapeutic treatment for the cervical region in the last three months
* Use of analgesics, anti-inflammatory drugs, or muscle relaxants in the last week; the presence of systemic diseases
* Medical diagnosis of fibromyalgia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2023-07-30 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Functional disability | Change from Baseline after 8 weeks of intervention and 4 weeks after the end of the intervention.
  The NDI will be used to verify the degree of disability due to neck pain.Each question has six potential responses ranging in severity from zero (no disability) to five (most severe disability) with a total score maximum of 50 points.
Numerical Pain Scale | Change from Baseline after 8 weeks of intervention and 4 weeks after the end of the intervention.
  The Numerical rating pain scale, a simple, easily administered scale evaluates the perceived intensity of pain, using an 11-point scale from 0, representing 'no pain', to 10, which is the 'worst possible pain'.

SECONDARY OUTCOMES:
Catastrophic Thoughts about Pain Scale | Change from Baseline after 8 weeks of intervention and 4 weeks after the end of the intervention.
  The Catastrophic Thoughts About Pain Scale will be used to assess pain-related catastrophizing. Thirteen items rated on 5 pont likert scales (0) not at all (4) all time. Higher score indicates higher level of Catastrophizing.
Kinesiophobia Tampa Scale | Change from Baseline after 8 weeks of intervention and 4 weeks after the end of the intervention.
  Tampa Kinesiophobia Scale will be used to assess fear of movement and injury recurrence. The TSK consists of 17 questions that assess fear of move- ment. The score for each item ranges from 1 to 4, where 1 represents ''strongly disagree'', 2 ''somewhat disagree'', 3 ''somewhat agree'', and 4 ''strongly agree''. For the final score, it is necessary to reverse the scores of questions 4, 8, 12, and 16. The total score varies between 17 and 68 points, and a higher score represents greater kinesiophobia.
The Copenhagen Neck Functional Disability Scale (CNFDS) | Change from Baseline after 8 weeks of intervention and 4 weeks after the end of the intervention.
  The CNFDS is a one-dimensional self-report scale consisting of 15 items that assess the degree of disability in activities of daily living in patients diagnosed with neck pain. When calculating the CNFDS score, the following procedures should be considered: For items 1 to 5, the answer "yes" = 0, "sometimes" = 1 and "no" = 2; For items 6 to 15, the answer "yes" = 2, "sometimes" = 1 and "no" = 0. Thus, the total score ranges from 0 to 30, the higher the score, the greater the disability.
Global Perception of Change scale | Change from Baseline after 8 weeks of intervention and 4 weeks after the end of the intervention.
  The perception of the global effect of the treatment by the research participant will be evaluated by the Global Perception of Change scale. The Global Perception of Change scale is a direct scale on the patient's self-perception when the intervention is performed. This scale consists of 11 points, ranging from -5 (worsening compared to the start of treatment), 0 (neutral) and +5 (improvement compared to the start of treatment), using the Portuguese version.

CONTACTS AND LOCATIONS:
Overall Officials: Cid Gomes, Phd, Principal Investigator — University of Nove de Julho
Locations (1):
- University of Nove de Julho, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Make data available remotely in digital cloud storage.

REFERENCES:
- [Derived] Barbosa da Silva AC, Santana GN, Santos IS, Dos Santos PG, de Oliveira AR, Filho AVD, de Paula Gomes CAF. Multimodal therapeutic intervention program associated with photobiomodulation therapy for individuals with chronic nonspecific neck pain: protocol for a clinical trial. Trials. 2024 Jul 3;25(1):442. doi: 10.1186/s13063-024-08289-1. PMID 38961460